CLINICAL TRIAL: NCT01535066
Title: Randomized Blinded Sham- and Waitlist-Controlled Trial of Acupuncture for Joint Symptoms Related to Aromatase Inhibitors in Women With Early Stage Breast Cancer
Brief Title: S1200: Acupuncture, Sham Acupuncture, or Wait List for Joint Symptoms Related to Aromatase Inhibitors in Pts W/Early-Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: S1200; S1200 (Other: SWOG); R01AT000636-01 (NIH); U10CA037429 (NIH); NCI-2012-00251 (Other: NCI)
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Pain
Keywords: estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; pain
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Experimental): Patients receive acupuncture therapy twice weekly for 6 weeks and then once weekly for 6 weeks.
  Interventions: Procedure: acupuncture therapy
- Arm II (Sham Comparator): Patients receive sham acupuncture twice weekly for 6 weeks and then once weekly for 6 weeks.
  Interventions: Procedure: sham acupuncture
- Arm III (No Intervention): Patients are assigned to a waiting list for 12 weeks with standard follow-up care.

INTERVENTIONS:
Procedure: acupuncture therapy — Receive acupuncture
  Arms: Arm I
Procedure: sham acupuncture — Receive sham acupuncture
  Arms: Arm II

SUMMARY:
RATIONALE: Acupuncture may help relieve joint pain.

PURPOSE: This randomized phase III trial studies acupuncture to see how well it works compared to sham acupuncture or waitlist in treating patients with joint pain related to aromatase inhibitors in patients with early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether true acupuncture administered twice weekly for 6 weeks (8-12 sessions) compared to sham acupuncture and waitlist control causes a significant reduction in joint pain related to aromatase inhibitors (AIs) in women with early-stage breast cancer as measured by the Brief Pain Inventory-Short Form (BPI-SF) worst pain score at 6 weeks.

Secondary

* To investigate the effects of true acupuncture administered twice weekly for 6 weeks (8-12 sessions) followed by 6 weekly treatments (4-6 sessions) of maintenance (12-18 sessions total over 12 weeks) compared to sham acupuncture and waitlist control in this study population; the evaluations at 12 and 24 weeks are to determine the benefit of additional 6 weekly acupuncture treatments for maintenance and to determine the durability of response after stopping acupuncture, respectively; the evaluation at 52 weeks is to determine the long-term effects of acupuncture and adherence to AIs.
* To evaluate the effects of acupuncture on the BPI-SF worst pain, worst stiffness, pain severity, and pain-related interference scores at 6, 12, 16, 20, 24, and 52 weeks.
* To evaluate the effects of acupuncture on Western Ontario and McMaster Universities Osteoarthritis (WOMAC) index (pain, stiffness, and function) for the hips and knees at 6, 12, 24, and 52 weeks.
* To evaluate the effects of acupuncture on Modified-Score for the Assessment and Quantification of Chronic Rheumatoid Affections of the Hands (M-SACRAH) (pain, stiffness, and function) at 6, 12, 24, and 52 weeks.
* To evaluate the effects of acupuncture on the PROMIS Pain Impact-Short Form (PROMIS PI-SF) at 6, 12, 24, and 52 weeks.
* To evaluate the effects of acupuncture on quality of life (QOL) as assessed by the Functional Assessment of Cancer Therapy-Endocrine Subscales (FACT-ES) at 6, 12, 24, and 52 weeks.
* To evaluate the effects of acupuncture on functional testing with grip strength and "Timed Get Up and Go" (TGUG) test at 6, 12, 24, and 52 weeks.
* To evaluate the effects of acupuncture on analgesic and opioid use at 2, 4, 6, 12, 16, 20, 24, and 52 weeks.
* To evaluate the effects of acupuncture on self-reported AI adherence at 12, 24, and 52 weeks.
* To assess AI adherence via urine AI metabolites at baseline, 24, and 52 weeks.
* To evaluate the effects of acupuncture on serum hormones (estradiol, FSH, LH) and inflammatory biomarkers (serum TNFα, IL-6, IL-12, CRP, and urine c-telopeptides of Type II collagen (CTX-II) at 6, 12, and 24 weeks. (Exploratory)
* To evaluate whether polymorphisms in CYP19A1 aromatase gene predict severity of AI-related joint symptoms. (Exploratory)
* To assess the safety and tolerability of acupuncture in this study population.

OUTLINE: This is a multicenter study. Patients are stratified according to study site. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive acupuncture twice weekly for 6 weeks and then once weekly for 6 weeks.
* Arm II: Patients receive sham acupuncture twice weekly for 6 weeks and then once weekly for 6 weeks.
* Arm III: Patients are assigned to a waiting list for 12 weeks. Patients complete the Brief Pain Inventory-Short Form (BPI-SF), the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index, the Modified-Score for the Assessment and Quantification of Chronic Rheumatoid Affections of the Hands (M-SACRAH), the PROMIS Pain Impact-Short Form (PROMIS PI-SF), the FACT-ES Trial Outcome Index, and the Aromatase Inhibitor Usage Form questionnaires at baseline and at 6, 12, 24 and 52 weeks.

Patients undergo blood sample collection at baseline and at 6, 12, and 24 weeks for serum hormones (estradiol, FSH, LH) levels, inflammatory markers (TNFα, IL-6, IL-12, CRP), and DNA analysis. Urine samples are also collected at baseline and at 24 and 52 weeks for c-telopeptides of Type II collagen and aromatase inhibitor metabolites analysis.

After completion of study treatment, patients are followed up at 24 and 52 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients must be women with histologically confirmed primary invasive carcinoma of the breast (Stage I, II, or III) with no evidence of metastatic disease (M0); patients must have undergone modified radical mastectomy or breast-sparing surgery; patients must have recovered from all side-effects of the surgery
* Patients must be positive for estrogen receptor (ER) and/or progesterone receptor (PgR) as determined by institutional standard
* Patients must currently be taking a third-generation aromatase inhibitor (AI) - anastrozole, letrozole, or exemestane for at least the previous 90 days prior to registration with plans to continue for at least an additional 1 year after registration; patients may have switched AIs provided that they have been on a stable dose for at least 90 days; concurrent trastuzumab (Herceptin) is allowed
* Patients must have completed the S1200 Brief Pain Inventory-Short Form (BPI-SF) within 14 days prior to registration; patients must have a worst pain score of at least 3 on the Brief Pain Inventory (item #2) that has started or increased since starting AI therapy
* Patients must be willing to submit blood and urine samples for serum hormones (estradiol, FSH, LH), inflammatory biomarkers (serum TNFα, IL-6, IL-12, CRP and urine CTX-II), urine AI metabolites, and DNA analysis (CYP19A1), and must be given the option to consent to use of remaining specimens for future translational medicine studies; baseline samples must be obtained prior to beginning intervention

PATIENT CHARACTERISTICS:

* Patients must be postmenopausal, as defined by at least one of the following:

  * ≥ 12 months since the last menstrual period
  * Prior bilateral oophorectomy
  * Current use of a gonadotropin-releasing hormone (GnRH) agonist
  * Previous hysterectomy with one or both ovaries left in place (or previous hysterectomy in which documentation of bilateral oophorectomy is unavailable) AND follicle-stimulating hormone (FSH) values consistent with the institutional normal values for the postmenopausal state; if patient is under the age of 55, FSH levels must be obtained within 28 days prior to registration
* Patients must have a Zubrod performance status of 0 to 1
* Patients must not have a severe bleeding disorder
* Patients must not have concurrent medical/arthritic disease that could confound or interfere with evaluation of pain or efficacy including: inflammatory arthritis (e.g., rheumatoid arthritis, systemic lupus, spondyloarthropathy, psoriatic arthritis, polymyalgia rheumatica), gout, episodes of acute monoarticular arthritis clinically consistent with pseudogout, Paget disease affecting the study joint (knees/hands), a history of septic arthritis or avascular necrosis or intra-articular fracture of the study joint, Wilson disease, hemochromatosis, alkaptonuria, or primary osteochondromatosis
* Patients must not have a history of bone fracture or surgery of the afflicted knees and/or hands within 6 months prior to registration
* Patients must not have a history of illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the patient
* Patients must be able to complete study questionnaires in English or Spanish
* No other prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, ductal carcinoma in situ [DCIS], adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer for which the patient has been disease-free for > 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Patients must not have had prior acupuncture treatment within the past 12 months or for AI-induced joint symptoms at any time
* Patients must not be on narcotics within 14 days of registration
* Patients must not have received oral corticosteroids, intramuscular corticosteroids, or intra-articular steroids within 28 days prior to registration
* Patients must not have received topical analgesics (e.g., capsaicin preparations) or any other analgesics (e.g., opiates or tramadol, with the exception of nonsteroidal anti-inflammatory drugs [NSAIDs] and acetaminophen) within 14 days prior to registration
* Patients must not have received or implemented any other medical therapy, alternative therapy, or physical therapy for the treatment of joint pain/stiffness within 28 days prior to registration; therapeutic massage is allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2012-05-16 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Decrease of joint pain associated with the use of AIs as measured by BPI-SF | 6 weeks

SECONDARY OUTCOMES:
Benefit of acupuncture maintenance as assessed by BPI-SF, WOMAC, M-SACRAH, PROMIS PI-SF, FACT-ES, and TGUG | 6, 12, 16, 20, and 24 weeks
Durability of response as assessed by BPI-SF, WOMAC, M-SACRAH, PROMIS PI-SF, FACT-ES, and TGUG | 52 weeks.
Long-term effects of acupuncture as assessed by BPI-SF, WOMAC, M-SACRAH, PROMIS PI-SF, FACT-ES, and TGUG | 52 weeks
Analgesic and opioid use | 2, 4, 6, 12, 16, 20, 24, and 52 weeks
AI adherence | 12, 24, and 52 weeks
Safety and tolerability of acupuncture | 2, 4, 6, 12, 16, 20, 24, and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, Principal Investigator — Herbert Irving Comprehensive Cancer Center
Locations (47):
- United States (47):
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente, Fremont, Fremont, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Columbia University Medical Center, New York, New York
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington

REFERENCES:
- [Derived] Hershman DL, Unger JM, Greenlee H, Capodice J, Lew DL, Darke A, Minasian LM, Fisch MJ, Henry NL, Crew KD. Comparison of Acupuncture vs Sham Acupuncture or Waiting List Control in the Treatment of Aromatase Inhibitor-Related Joint Pain: A Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2241720. doi: 10.1001/jamanetworkopen.2022.41720. PMID 36367721
- [Derived] Hershman DL, Unger JM, Greenlee H, Capodice JL, Lew DL, Darke AK, Kengla AT, Melnik MK, Jorgensen CW, Kreisle WH, Minasian LM, Fisch MJ, Henry NL, Crew KD. Effect of Acupuncture vs Sham Acupuncture or Waitlist Control on Joint Pain Related to Aromatase Inhibitors Among Women With Early-Stage Breast Cancer: A Randomized Clinical Trial. JAMA. 2018 Jul 10;320(2):167-176. doi: 10.1001/jama.2018.8907. PMID 29998338
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/